CLINICAL TRIAL: NCT05803850
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Doses (SAD) Study Following Oral Administration in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of HNC1058
Brief Title: A Study to Evaluate the Safety, Tolerability, PK and PD of HNC1058
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Henovcom Bioscience Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HNC1058-A101
Record Dates: First submitted 2023-03-23; First posted 2023-04-07 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: IPF

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HNC1058 Capsules (Experimental): HNC1058 Capsules, single ascending doses
  Interventions: Drug: HNC1058 Capsules
- HNC1058 Placebos (Placebo Comparator): HNC1058 Placebos, single ascending doses
  Interventions: Drug: HNC1058 Capsules
- HNC1058 Capsules FED (Experimental): HNC1058 Capsules, food effect, Single dose
  Interventions: Drug: HNC1058 Capsules
- HNC1058 Placebos FED (Placebo Comparator): HNC1058 Placebos, food effect, Single dose
  Interventions: Drug: HNC1058 Capsules

INTERVENTIONS:
Drug: HNC1058 Capsules — HNC1058 Capsules/Placebos, single dose, PO, starting dose of 10 mg escalating up to 80 mg；HNC1058 Capsules/Placebos, 50 mg, single dose, FED.
  Other Names: HNC1058 Placebos

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety and tolerability after single ascending oral doses of HNC1058 given to healthy subjects, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent; willing and able to comply with the schedule, requirements, and restrictions of the study. Are capable of giving informed consent and complying with study procedures.
2. Between the ages of 18 and 55 years (inclusive) at the time of Screening.
3. BMI between 18.0 and 32.0 kg/m2 (inclusive) at the time of Screening and have a body weight no less than 50 kg.
4. In good general health, as determined by the Investigator.
5. Female subjects must be non pregnant and non lactating.
6. Female subjects must be of non childbearing potential, or agree to use an appropriate method(s) of contraception throughout the entire duration of study participation, and have negative pregnancy test results at Screening (serum) and Admission (urine).

   Refer to Section 6.4.1 for full details of reproductive requirements and acceptable methods of contraception for female subjects.
7. Male subjects with female partners of reproductive potential must agree to practice abstinence or to use a condom (male subject) plus an additional barrier method (female partner) of contraception for the duration of the study and for at least 90 days after dosing; must also agree to refrain from sperm donation for at least 90 days post dose.
8. Normal renal function as determined by Investigator following review of clinical laboratory test results, including eGFR as estimated using the CKD EPI equation.
9. Non smoker, with no use of any tobacco or nicotine containing products within 6 months prior to Day 1.

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator.
2. Known or suspected malignancy.
3. History of pancreatitis or gall stones.
4. History of unexplained syncope, symptomatic hypotension, or hypoglycemia.
5. Family history of long QTc syndrome.
6. History of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance.
7. Poor venous access.
8. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B, hepatitis C, or hepatitis E.
9. Hospital admission or major surgery within 6 months prior to screening.
10. History of alcohol or prescription drug abuse within 9 months prior to screening.
11. Positive test result for alcohol or drugs of abuse (i.e., UDS) at screening or Admission.
12. Use of any prohibited medication(s) and/or substance(s), including:

    1. use of any drugs known to induce or inhibit drug metabolism within 30 days prior to Day 1;
    2. receipt of another investigational medication (EXCEPT biological compound) within 30 days or receipt of biological compound within 90 days (or 5 half lives, whichever is longer) prior to Day 1;
    3. participation in an investigational device study within 30 days prior to Day 1.
    4. routine consumption of the following within 14 days prior to Day 1:

    i. Prescription medication (except hormonal contraception for WOCBP), OTC medication, traditional Chinese medicine, or herbal medicine (within 14 days or 5 half lives, whichever is longer); ii. Vitamin, mineral, and other dietary supplements; iii. Grapefruit and grapefruit juice; e. donation of the following within the below specified timeframe prior to Day 1: i. bone marrow or peripheral stem cells within 90 days; ii. blood within 60 days; iii. plasma within 30 days. f. Any of the following activities within 72 hours prior to Day 1: i. strenuous exercise; ii. alcohol consumption; iii. consumption of caffeine-containing substances.
13. Loss of >500 mL blood (for any reason) within 90 days prior to Day 1.
14. For 50 mg cohort only: inability to completely consume a standardized high fat breakfast within 30 minutes.
15. Per investigator discretion, any other reason that would render a subject inappropriate for study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and concomitant medications | Between screening and 7-9 days after the last dose
  To evaluate the safety and tolerability of HNC1058 in comparison with placebo after a single oral dose in healthy subjects in terms of AEs and CMs.

SECONDARY OUTCOMES:
Number of subjects with vital sign measurements | Between screening and 7-9 days after the last dose
  To evaluate the safety and tolerability of HNC1058 in comparison with placebo after a single oral dose in healthy subjects in terms of abnormal vital signs
Number of subjects with clinical laboratory test results | Between screening and 7-9 days after the last dose
  o evaluate the safety and tolerability of HNC1058 in comparison with placebo after a single oral dose in healthy subjects in terms of abnormal clinical laboratory test results

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No